CLINICAL TRIAL: NCT02571270
Title: Impact Of Supervised 12-Week-Combined Physical Training In Heart Failure Patients: A Randomized Trial
Brief Title: 12-Week-Combined Physical Training In Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Tainá Fabri, Master's degree, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UEPJMF-001
Record Dates: First submitted 2015-10-02; First posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure Patients
Keywords: Exercise; quality of life; healthy; cardiac remodeling
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- Active lifestyle (Active Comparator): Active lifestyle involves nutritional education, physical activity and active recreation.
  Interventions: Other: Combined aerobic and resistance physical training program
- Lifestyle counseling (Active Comparator): Lifestyle counseling helps patients to have better self-care.
  Interventions: Other: Combined aerobic and resistance physical training program
- secondary prevention (Active Comparator): Secondary prevention it is essential to prevent a new unfavorable event.
  Interventions: Other: Combined aerobic and resistance physical training program
- survival (Active Comparator): The survival of patients with heart failure may increase with exercise training.
  Interventions: Other: Combined aerobic and resistance physical training program

INTERVENTIONS:
Other: Combined aerobic and resistance physical training program

SUMMARY:
Purpose: Physical exercise exerts favorable impact on functional capacity (FC) and quality of life (QL) in patients with heart failure (HF). It is believed that the combined aerobic and resistance physical training (CPT) supervised by physical educator is better than only prescription of unsupervised exercise. The aim of this study is to compare the effects of a CPT program on the FC and QL of HF patients with reduced ejection fraction (HFREF) with the practice medical routine prescription of regular physical activity and correlate these findings with clinical and echocardiographic variables.

Methods: A longitudinal prospective study included 28 consecutive HFREF patients randomly divided in two age- and gender- matched groups: Trained Group (TG, n = 17), patients undergoing 12 weeks of supervised CPT and Non Trained Group (NTG, n = 11), patients receiving only medical prescription to practice regular physical exercise. All patients were submitted to clinical evaluation, transthoracic echocardiography, Cooper walk test and QL questionnaire before and after the study protocol. Student t test or Mann-Whitney test were performed for groups comparison and correlation tests for the same group variable associations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure with LVEF <50%;
* Patients with optimized drug therapy;
* Age over 18 years.

Exclusion Criteria:

* Heart failure NYHA class IV and/or Stage D;
* Decompensated HF in the last three months;
* Atrial fibrillation and/or implantable device at the moment of inclusion;
* Patients with chronic obstructive pulmonary disease (COPD);
* Patients with biomechanical limitations of physical activity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Questionnaire about quality of life | up to 12 weeks of research
Cardiorespiratory evaluation (VO2 in Mets) | up to 12 weeks of research
Morphological echocardiographic variables (mm) | up to 12 weeks of research
Sistolic Function echocardiographic variables (Percentage) | up to 12 weeks of research
Diastolic Function echocardiographic variables (cm/s) | up to 12 weeks of research

SECONDARY OUTCOMES:
Anthropometric measurements (cm) | up to 12 weeks of research
Body composition (%fat percentage) | up to 12 weeks of research
Presence of comorbidities | up to 12 weeks of research
Blood pressure measurement (mmHg) | up to 12 weeks of research